CLINICAL TRIAL: NCT04422717
Title: Ultrasonographic Evaluation of Femoral Cartilage Thickness In Patients With Lower Limb Amputation
Brief Title: Femoral Cartilage Thickness In Patients With Lower Limb Amputation
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstanbulPMRTRH-HCK1
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Amputation; Osteo Arthritis Knee
Keywords: Amputate; rehabilitation; ultrasonography; osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study to investigate any relation with functional parameters and femoral cartilage thickness evaluation by ultrasonography in lower extremity amputate individuals.

DETAILED DESCRIPTION:
In this prospective observational study, subjects approached Tertiary Rehabilitation Clinics for prothesis recipe or long term outpatient follow up was 150 people. Among them 76 subjects accepted to enroll study. Informed consent was taken. Subjects firstly performed clinical parameters at the first doctor's control. Knee radiography has been performed.

ELIGIBILITY:
Inclusion Criteria:

* Being a single lower limb amputation
* At least one year after the amputation operation
* Prosthesis use for the last 6 months
* Being traumatic or vascular
* Not having stump infection
* Muscle strength over stump should be at least 3/5

Exclusion Criteria:

* Doing quadriceps exercise in the last 3 months
* Trauma, surgery, and knee injections within 6 months (PRP, hyaluronic acid), Chondroitin-glucosamine use.

Being any of the active synovitides, Rheumatoid arthritis, spondyloarthritis, pseudogout, coxarthrosis, neuromuscular diseases

* Having an additional disease that will cause psychiatric adjustment problem
* Subjects are younger than 18 years
* Bilateral amputated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective observational study, subjects approached Tertiary Rehabilitation Clinics for prothesis recipe or long term outpatient follow up was 150 people. Among them 76 subjects accepted to enroll study.İnformed consent was taken.1 subject not acceptable with inclusion criteria was excluded.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Evaluation of Femoral Cartilage Thickness | Day 1
  The transtibial amputee's both knees femoral cartilage are measured. The transfemoral group is measured only femoral cartilage of intact side. 10 subjects are randomised for intraobserver reliability and reevaluated one month after their first measure.

SECONDARY OUTCOMES:
Trinity Amputation and Prosthesis Experience Scale (TAPES) | Day 1
  Trinity Amputation and Prosthesis Experience Scale(3 parts) TAPES Psychosocial maximum:75 minimum:15 points. Higher points indicate better psychosocial outcomes. TAPES activity restriction Maximum:24 minimum:0 points. Higher points indicate more activity restricted. TAPES Prosthesis Pleasant Maximum:75 Minimum:15 higher points indicate much pleasant about prothesis
Houghton Scale | Day 1
  The Houghton scale is a 4-item instrument that accesses prosthetic use in people with lower extremity amputations. It reflects a person's perception of prosthetic use. It's self-administered and easy to score. Maximum:12 points. Minimum:0 Higher scores indicate better accesses.
Short Form - 12 (SF-12) | Day 1
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. Maximum:43 points minimum:12 points. Higher points indicate a higher quality of life.
Falls Efficacy Scale | Day 1
  On a scale from 1 to 10, with 1 being very confident and 10 being not confident at all, how confident are you that you do the following activities without falling? A total score of greater than 70 indicates that the person has a fear of falling. Minimum:0 Maximum:100 points.
Medicare Functional Classification Levels (K levels) | Day 1
  Level 0: Does not have the ability or potential to ambulate or transfer safely with or without assistance and a prosthesis does not enhance their quality of life or mobility Level 1: Has the ability or potential to use a prosthesis for transfers or ambulation on level surfaces at fixed cadence. Typical of the limited and unlimited household ambulators.
  Level 2: Has the ability or potential for ambulation with the ability to traverse low-level environmental barriers such as curbs, stairs, or uneven surfaces. Typical of the limited community ambulator.
  Level 3: Has the ability or potential for ambulation with variable cadence. Typical of the community ambulator who has the ability to traverse most environmental barriers and may have vocational, therapeutic, or exercise activity that demands prosthetic utilization beyond simple locomotion.
  Level 4: Typical of the prosthetic demands of the child, active adult, or athlete. Minimum: K0 Maximum: K4
Locomotor Capabilities Index (LCI) -5 | Day 1
  The LCI is a disease-specific, self-administered instrument for assessing locomotor abilities generally considered essential for basic and advanced activity daily livings of people with lower-limb amputation and an enabling factor associated with long-term prosthetic use. It is easily administered and quickly completed. Maximum:56 Minimum:0 points. Higher scores indicate better locomotor capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Habip Can Küçük, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akkaya N, Akkaya S, Ozcakar L, Demirkan F, Kiter E, Konukcu S, Ardic F. Ultrasonographic measurement of the distal femoral cartilage thickness in patients with unilateral transtibial amputation. Prosthet Orthot Int. 2013 Aug;37(4):268-74. doi: 10.1177/0309364612464233. Epub 2012 Nov 9. PMID 23144161
- [Result] Kesikburun S, Koroglu O, Yasar E, Guzelkucuk U, Yazcoglu K, Tan AK. Comparison of Intact Knee Cartilage Thickness in Patients with Traumatic Lower Extremity Amputation and Nonimpaired Individuals. Am J Phys Med Rehabil. 2015 Aug;94(8):602-8. doi: 10.1097/PHM.0000000000000216. PMID 25299529
- [Result] Sahin Onat S, Malas FU, Ozturk GT, Akkaya N, Kara M, Ozcakar L. Ultrasonographic assessment of the quadriceps muscle and femoral cartilage in transtibial amputees using different prostheses. Prosthet Orthot Int. 2016 Aug;40(4):484-9. doi: 10.1177/0309364615592701. Epub 2015 Jul 9. PMID 26163535
- [Result] Ozcakar L, Tunc H, Oken O, Unlu Z, Durmus B, Baysal O, Altay Z, Tok F, Akkaya N, Dogu B, Capkin E, Bardak A, Carli AB, Bugdayci D, Toktas H, Diracoglu D, Gunduz B, Erhan B, Kocabas H, Erden G, Gunendi Z, Kesikburun S, Omac OK, Taskaynatan MA, Senel K, Ugur M, Yalcinkaya EY, Ones K, Atan C, Akgun K, Bilgici A, Kuru O, Ozgocmen S. Femoral cartilage thickness measurements in healthy individuals: learning, practicing and publishing with TURK-MUSCULUS. J Back Musculoskelet Rehabil. 2014;27(2):117-24. doi: 10.3233/BMR-130441. PMID 24284270